CLINICAL TRIAL: NCT02155088
Title: A Phase I Trial With Cohort Expansion of BYL719 in Combination With Gemcitabine and (Nab)-Paclitaxel in Locally Advanced and Metastatic Pancreatic Cancer
Brief Title: BYL719 in Combination With Gemcitabine and (Nab)-Paclitaxel in Locally Advanced and Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17815
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Cancer
Keywords: Locally Advanced; Metastatic; Recurrent; Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Alpelisib; Gemcitabine; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy: BYL719, Gemcitabine, (Nab)-Paciltaxel (Experimental): Dose escalation, followed by expansion, of BYL719 in combination with Gemcitabine and (Nab)-Paclitaxel. BYL719: once daily. Gemcitabine: Days 1,8, 15 of 28-day cycle. (Nab)-Paclitaxel: Days 1,8, 15 of 28-day cycle.
  Interventions: Drug: BYL719; Drug: Gemcitabine; Drug: (nab)-paclitaxel

INTERVENTIONS:
Drug: BYL719 — Dose escalation beginning at 250 mg/day
  Other Names: a-specific P13K inhibitor
Drug: Gemcitabine — Dose escalation beginning at 800 mg/m^2
  Other Names: Gemzar
Drug: (nab)-paclitaxel — 125 mg/m^2 dose
  Other Names: Abraxane

SUMMARY:
The main purpose of this study is to see primarily if BYL719 is safe to be given to patients in combination with gemcitabine and nab-paclitaxel. Gemcitabine and nab-paclitaxel is an FDA-approved regimen to treat pancreatic cancer. Secondary goals will be to find out the effect on tumor of this new drug combination of BYL719, gemcitabine and nab-paclitaxel. In the first part of the study, different doses of BYL719 will be tested. In the second part of the study, all patients will be started at the same dose of BYL719.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to swallow and retain oral medication
* Histologically documented diagnosis of pancreatic adenocarcinoma.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Required baseline laboratory status according to protocol document

Exclusion Criteria:

* Prior sensitivity or intolerance to PI3K inhibitors
* Potential participants with central nervous system (CNS) involvement may participate if the patient is: >/= 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment; Clinically stable with respect to the CNS tumor at the time of screening; Not receiving steroid therapy.
* Prior treatment with any cytotoxic chemotherapy for treatment of pancreatic cancer except as an adjuvant therapy. Should not have received gemcitabine within 6 months of starting the study treatment. 5-Fluorouracil or radiation treatment should be received more than 4 weeks prior to receiving the study drug.
* Potential participants who have received radiotherapy ≤ 4 weeks prior to starting study drugs, with exception of palliative radiotherapy, who have not recovered from side effects of such therapy to baseline or Grade ≤ 1 and/or from whom ≥ 30% of the bone marrow was irradiated.
* Potential participants who have undergone major surgery ≤ 4 weeks prior to starting study treatment or who have not recovered from side effects of such procedure.
* Have received investigation agent within 30 days prior to enrollment
* Clinically significant cardiac disease or impaired cardiac function
* QT interval adjusted according to Fredericia (QTcF) > 480 msec on screening ECG
* Potential participants with diabetes mellitus requiring insulin treatment and/or with clinical signs or with fasting plasma glucose (FPG)> 140 mg/dL or history of documented steroid-induced diabetes mellitus.
* Any other condition that would, in the Investigator's judgment, preclude participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g. infection/inflammation, intestinal obstruction, unable to swallow oral medication, social/psychological complications.
* Impaired GI function or GI disease that may significantly alter the absorption of oral BYL719 (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable hepatitis B virus [HBV]-DNA and/or positive HbsAg, quantifiable hepatitis C virus [HCV]-RNA).
* Known positive serology for human immunodeficiency virus (HIV)
* Known severely impaired lung function (spirometry and diffusing capacity of lung for carbon monoxide[DLCO] 50% or less of normal and O2 saturation 88% or less at rest on room air).
* Currently receiving warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed
* Currently receiving treatment with drugs known to be strong inhibitors or inducers of isoenzyme CYP3A. Must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the start of treatment. Switching to a different medication prior to starting study treatment is allowed.
* Has a history of non-compliance to medical regimen or inability to grant consent
* Currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (TdP) and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug treatment
* History of another malignancy requiring active treatment within 2 years prior to starting study treatment, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 5 mIU/mL)
* Participant who does not apply highly effective contraception during the study and through 12 weeks after final dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 4 months per participant
  The MTD is defined as the highest dose level at which one or none of 6 patients experience a Dose Limiting Toxicity (DLT).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 3 years
  Complete Response plus Partial Response (CR+PR). CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Overall Survival (OS) | Up to 3 years
  Overall survival of patients who receive at least one dose of the study drug at MTD.
Progression-Free Survival (PFS) | Up to 3 years
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States